CLINICAL TRIAL: NCT04676204
Title: STATURE: A Prospective Observational Study of the relationShip beTween Oral DMT bURden and adhErence in People With MS
Brief Title: Relationship Between Oral DMT Burden and Adherence in MS
Acronym: STATURE
Status: Enrolling by invitation | Type: Observational
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Ernest Butler, Principle Investigator, Monash University
Other Study IDs: STATURE01
Record Dates: First submitted 2020-11-25; First posted 2020-12-19 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis; Adherence, Medication
Keywords: Multiple Sclerosis; Adherence; Treatment Burden; Disease Modifying Therapy; Oral; Cladribine; Dimethyl fumarate; Fingolimod; Teriflunomide; Ozanimod; Diroximel Fumarate
MeSH Terms: conditions — Multiple Sclerosis; Medication Adherence | interventions — Cladribine; Dimethyl Fumarate; Fingolimod Hydrochloride; teriflunomide; ozanimod; diroximel fumarate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cladribine: Participants with MS commencing cladribine disease modifying treatment as clinically prescribed.
  Interventions: Drug: Cladribine
- Dimethyl Fumarate: Participants with MS commencing dimethyl fumarate disease modifying treatment as clinically prescribed.
  Interventions: Drug: Dimethyl fumarate
- Fingolimod: Participants with MS commencing fingolimod disease modifying treatment as clinically prescribed.
  Interventions: Drug: Fingolimod
- Teriflunomide: Participants with MS commencing teriflunomide disease modifying treatment as clinically prescribed.
  Interventions: Drug: Teriflunomide
- Ozanimod: Participants with MS commencing Ozanimod disease modifying treatment as clinically prescribed.
  Interventions: Drug: Ozanimod
- Diroximel Fumarate: Participants with MS commencing diroximel fumarate disease modifying treatment as clinically prescribed.
  Interventions: Drug: Diroximel fumarate

INTERVENTIONS:
Drug: Cladribine — Cladribine is a purine antimetabolite indicated for the treatment of relapsing forms of multiple sclerosis, to include relapsing-remitting disease and active secondary progressive disease, in adults.
  Other Names: Mavenclad
  Groups: Cladribine
Drug: Dimethyl fumarate — Dimethyl fumarate is indicated for the treatment of relapsing forms of multiple sclerosis, to include clinically isolated syndrome, relapsing-remitting disease, and active secondary progressive disease, in adults
  Other Names: Tecfidera
  Groups: Dimethyl Fumarate
Drug: Fingolimod — Fingolimod is a sphingosine 1-phosphate receptor modulator indicated for the treatment of patients with relapsing forms of multiple sclerosis to reduce the frequency of clinical exacerbations and to delay the accumulation of physical disability.
  Other Names: Gilenya
  Groups: Fingolimod
Drug: Teriflunomide — Teriflunomide is a pyrimidine synthesis inhibitor indicated for the treatment of patients with relapsing forms of multiple sclerosis.
  Other Names: Aubagio
  Groups: Teriflunomide
Drug: Ozanimod — Ozanimod is a sphingosine-1-phosphate receptor modulator indicated for the treatment of patients with relapsing forms of multiple sclerosis.
  Other Names: Zeposia
  Groups: Ozanimod
Drug: Diroximel fumarate — Diroximel fumarate is indicated for the treatment of relapsing forms of multiple sclerosis, to include clinically isolated syndrome, relapsing-remitting disease, and active secondary progressive disease, in adults.
  Other Names: Vumerity
  Groups: Diroximel Fumarate

SUMMARY:
STATURE is a prospective observational six-arm translation multi-site study that will run for approx. 4.5 years. The primary aim is to measure treatment burden and its relationship to medication adherence across six self-administered oral disease-modifying therapies (cladribine, dimethyl fumarate, fingolimod, teriflunomide, ozanimod, and diroximel fumarate) in multiple sclerosis (MS). The information gained will assist prescribing decision-making; accounting for medication burden at a patient level and potential implications on medication adherence and persistence, thus minimising primary and secondary healthcare costs. Three-hundred and twenty-three individuals with MS will be recruited into the study. Patient-reported outcome measures will be administered via Qualtrics, a secure online data collection tool. Medicare and pharmaceutical benefits scheme (PBS) data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* A confirmed diagnosis of multiple sclerosis.
* Commencement (switching or newly prescribed) of one of the 6 following DMTs within the previous 2-months: cladribine, dimethyl fumarate, fingolimod, teriflunomide, ozanimod, diroximel fumarate.
* Able to read and write in English.
* Access to an internet connection and computer facilities, required to complete assessments.

Exclusion Criteria:

* Use of any other DMT than cladribine, dimethyl fumarate, fingolimod, teriflunomide, ozanimod, diroximel fumarate.
* Comorbid neurological condition.
* Severe cognitive or psychological dysfunction deemed to interfere with the person's ability to undertake study requirements, as determined by their MS clinic treatment team (neurologist; MS nurse).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three-hundred and twenty-three people with MS, who have recently commenced (<2-months) one of the six oral DMTs under investigation during routine clinical care
Sampling Method: Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-11-19 (Estimated); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
Medication Burden | 24-months
  Identification of medication burden will be calculated into indices of pre-workup and monitoring time, refill and administration and side-effects. This will allow the development of an indices of overall perceived burden, as well as sub-indices of specific perceived burden.
Medication Adherence (MPR) | 24-months
  Identification of medication adherence, persistence and switching between oral DMTs will be calculated as the medication possession ratio (MPR) collected from pharmaceutical benefit scheme claims over the 24-month enrollment period. In addition, basic self-reported adherence and discontinuation will be collected.
Medication Adherence (PDC) | 24-months
  Identification of medication adherence, persistence and switching between oral DMTs will be calculated as the proportion of days covered (PDC) collected from pharmaceutical benefit scheme claims over the 24-month enrollment period. In addition, basic self-reported adherence and discontinuation will be collected.

SECONDARY OUTCOMES:
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | 24-Months
  The Multiple Sclerosis Quality of Life-54 (MSQOL-54) is a structured, self-report questionnaire examining quality of life that contains 54-items, generating 12 subscales with two summary scores (physical health and mental health) and two additional single-item measures (satisfaction with sexual function and change in health). In scoring the MSQOL-54, two summary scores (physical and mental health) are produced from a weighted combination of scale scores, where scale scores range from 0 to 100, with higher scale score indicating improved quality of life. Quality of life (QoL) is being utilised as an outcome measure to identify whether QoL is predicted by 24-month MPR/PDC adherence and persistence.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Butler, PhD; MD, Principal Investigator — Monash University; Monash Health
Locations (1):
- Monash University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT04676204/ICF_000.pdf